CLINICAL TRIAL: NCT00400686
Title: A Single Institution, Open-Label, Nonrandomized Pilot Study of High Dose Epoetin Alfa Administered Once a Week in Patients With Multiple Myeloma: Its Effects on Hemoglobin, Blood Transfusion Requirements and Quality of Life
Brief Title: Epoetin Alfa in Treating Anemia in Patients Undergoing Chemotherapy for Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE-CCF-5497; P30CA043703 (NIH); CASE-CCF-5497 (Other: Cleveland Clinic); ORTHO-CASE-CCF-5497 (Other: Cleveland Clinic)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Anemia; Multiple Myeloma; Plasma Cell Neoplasm
Keywords: anemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Anemia; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epoetin Alfa - 80,000 U sc (Experimental): Epoetin Alfa will be administered 80,000 units subcutaneously every week beginning on Day 1. On Day 28, the dose was adjusted based upon patients' Hemoglobin Levels
  Interventions: Biological: epoetin alfa

INTERVENTIONS:
Biological: epoetin alfa — Epoetin alfa will be administered 80,000 u sc every week commencing on study day 1.

SUMMARY:
RATIONALE: Epoetin alfa may cause the body to make more red blood cells. It is used to treat anemia in patients with multiple myeloma.

PURPOSE: This clinical trial is studying how well epoetin alfa works in treating anemia in patients undergoing chemotherapy for multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the hematologic response and transfusion requirements of chemotherapy-related moderate anemia to the administration of a high initial dose of epoetin alfa followed by a less frequent maintenance dose of epoetin alfa in multiple myeloma patients.

Secondary

* Determine the effect of moderate anemia on quality of life in these patients.
* Correlate changes in hemoglobin levels with changes in quality of life in patients treated with this drug.
* Determine the effect of this drug on transfusion requirements after day 28 in these patients.

OUTLINE: This is an open-label, non-randomized, pilot study.

Patients receive high-dose epoetin alfa subcutaneously (SC) once a week for 4 weeks or until their hemoglobin levels reach 12-13 g/dL. Patients then receive epoetin alfa SC once every 2 weeks for 8 weeks OR once a week for 4 weeks, and then once every 2 weeks for 8 weeks (as long as their hemoglobin levels remain between 12-13 g/dL). Patients then receive maintenance epoetin alfa SC once every 4 weeks for up to 12 weeks.

Patients whose hemoglobin level decreases by 1-1.5 g/dL return to previous epoetin alfa schedule. Patients whose hemoglobin level is < 9 g/dL after returning to the previous schedule may receive epoetin alfa for an additional 24 weeks.

Quality of life is assessed at baseline and at weeks 2, 4, 8, 16, and 24 weeks during treatment.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma (MM)
* Requiring active therapy for MM

  * Planning to undergo chemotherapy for ≥ 3 months
* Moderate anemia caused by MM and/or chemotherapy, as evidenced by hemoglobin ≤ 11.0 g/dL
* No untreated anemia predominantly due to factors other than MM/chemotherapy (i.e., iron or folate deficiencies, hemolysis, HIV, or gastrointestinal bleeding)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Life expectancy ≥ 6 months
* Transferrin saturation ≥ 20%
* Ferritin ≥ 100 ng/mL
* Homocysteine normal (concurrent vitamin supplementation allowed)
* Methylmalonic acid normal (concurrent vitamin supplementation allowed)
* Renal function normal
* No uncontrolled hypertension
* No prior thrombotic events unless treated with appropriate prophylaxis
* No known hypersensitivity to mammalian cell-derived products
* No uncontrolled infection
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight < 100 Kg
* Patients with iron, folate, or vitamin B_12 deficiency allowed provided conditions are corrected prior to study entry
* Able to read and understand English at a 7th grade level

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior total lymphoid, extensive abdominal, or inverted Y radiotherapy
* Concurrent red blood cell transfusion allowed provided hemoglobin ≤ 7 g/dL AND patient is symptomatic
* Concurrent vitamin supplementation allowed for cyanocobalamin (vitamin B_12) or folate deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-09; Primary Completion 2009-01 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Sobecks, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 9/2003 to 6/2008, a total of 31 patients were enrolled.
Period: Overall Study
Arm/Group | Epoetin Alfa - 80,000 U sc
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epoetin Alfa - 80,000 U sc
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 61.9 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin at Day 28
Description: Change from baseline in hemoglobin after treatment with high-dose Epoetin Alfa.
Time Frame: Baseline to Day 28
Measure: Median (Full Range); unit: g/dL
Arm/Group | Epoetin Alfa - 80,000 U sc
Number analyzed (Participants) | 31
g/dL | 1.3 [-3.0 to 4.4]

2. Primary Outcome: Number of Patients With an at Least 1gm/dL Increase in Hgb
Time Frame: Baseline to Day 28
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa - 80,000 U sc
Number analyzed (Participants) | 31
participants | 13

3. Primary Outcome: Number of Patients With an at Least 2gm/dL Increase in Hgb
Time Frame: Baseline to Day 28
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa - 80,000 U sc
Number analyzed (Participants) | 31
participants | 9

ADVERSE EVENTS:
Time Frame: AE data highlights development of VTEs in patients receiving one of the following: 1. lenalidomide, high dose dexamethasone & Aspirin 325mg daily 2. thalidomide & doxil based therapy with aspirin 81mg daily 3. cyclophosphamide & prednisone without VTE
Description: Only immediately reportable Serious Adverse Events (SAE) & Venous thrombolytic event (VTE) were captured for the purpose of this study.
Arm/Group | Epoetin Alfa - 80,000 U sc
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 3/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoetin Alfa - 80,000 U sc (N=31)
Venous Thromboembolic Event (VTE) (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No